CLINICAL TRIAL: NCT03048981
Title: Effects of Fish Oil on Platelet Function and Coagulation
Acronym: FOILP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Thomas Kander, Principal investigator, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Fish oil and platelet function
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Platelet Aggregation, Spontaneous; Atherosclerosis; Surgery
Keywords: Thrombocyte aggregation; Fish oil; Alternative medicine; Point of care testing; Coagulation monitoring
MeSH Terms: conditions — Platelet Aggregation, Spontaneous; Atherosclerosis | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Before and after
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fish oil intake (Experimental): Healthy volunteers given maximum dose of fish oil for 10 days.
  Interventions: Drug: Fish oil

INTERVENTIONS:
Drug: Fish oil — Blood samples before and after 10 day intake of maximum dose fish oil

SUMMARY:
Many patients undergoing surgery use naturopathic drugs, including fish oil. Fish oil has been reported to increase bleeding in patients through inhibiting platelet aggregation and prolonging of clot formation time. The Swedish Medical Products Agency recommends that patients stop taking the naturopathic medicines including fish oil two weeks prior planed surgery. The aim of this study is to examine the effects of fish oil given to healthy volunteers using point of care coagulation assessment and flow dependent Cellix instrument before and after intake of fish oil.

DETAILED DESCRIPTION:
Healthy volunteers will be given maximum dose of fish oil for 7 days. Blood samples will be collected before and immediately after the 7 days of intake and analysed using point of care coagulation assessment instruments and flow dependent platelet aggregation using a microfluid flow controlled system (Cellix). For point of care coagulation assessment the multiple electrode platelet aggregometer Multiplate, the viscoelastic rotational thromboelastometers ROTEM and Sonoclot will be used. Flow cytometry may also be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking healthy volunteers with written consent to participate

Exclusion Criteria:

* Medication affecting coagulation or platelets within 14 days priori to inclusion

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Thrombocyte aggregation measured with multiple electrode aggregometry | Change of thrombocyte aggregation directly after intake period of 7 days compared to baseline
  Multiple electrode aggregometry gives a area under the curve proportional to thrombocyte aggregation
Thrombocyte aggregation measured with Cellix's microfluidic pumps and biochips | Change of thrombocyte aggregation directly after intake period of 7 days compared to baseline
  Cellix's microfluidic pumps and biochips gives an thrombosis area proportional to thrombocyte aggregation

SECONDARY OUTCOMES:
Coagulation measured with the viscohemostatic instrument ROTEM | Change of coagulation directly after intake period of 7 days compared to baseline
  Viscohemostatic instrument
Coagulation measured with the viscohemostatic instrument and Sonoclot | Change of coagulation directly after intake period of 7 days compared to baseline
  Viscohemostatic instrument

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, MD, Phd, Principal Investigator — Dept. of Clinical Sciences, Lund University, SWEDEN
Locations (1):
- Intensive and perioperative care. Skåne University Hospital. Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon reasonable request

REFERENCES:
- [Result] Bagge A, Schott U, Kander T. Effects of naturopathic medicines on Multiplate and ROTEM: a prospective experimental pilot study in healthy volunteers. BMC Complement Altern Med. 2016 Feb 17;16:64. doi: 10.1186/s12906-016-1051-y. PMID 26887420